CLINICAL TRIAL: NCT00547560
Title: An Ascending Multiple Dose Study Of The Safety, Pharmacokinetics, And Pharmacodynamics Of GSI-953 Administered Orally To Healthy Elderly Subjects
Brief Title: Study Evaluating Multiple Doses Of GSI-953 Within The Elderly Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3183A1-102; B1941003
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — begacestat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GSI+Placebo (Other)
  Interventions: Drug: GSI-953

INTERVENTIONS:
Drug: GSI-953 — Oral capsule, 10- and 50-mg, either once a day for 14 days or twice a day for 14 days, depending on cohort assignment.
  Other Names: Begacestat, WAY-210953, PF-05212362

SUMMARY:
To assess the safety and tolerability of ascending, multiple, oral doses of GSI-953 in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, greater than or equal to 65 years of age.
* Women of nonchildbearing potential (WONCP) may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for greater than or equal to 1 year (with FSH greater than or equal to 38 mIU/mL) and must have a negative pregnancy test result within 48 hours before administration of test article. Women who are surgically sterile must provide documentation of the procedure by an operative report or by ultrasound.
* Body mass index (BMI) in the range of 18.0 to 30.0 kg/m2 and body weight >50 kg.

Exclusion Criteria:

n/a

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic and pharmacodynamic profile for the elderly subjects. | 6 months

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | 6 months
Pharmacodynamics (PD) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3183A1-102&StudyName=Study%20Evaluating%20Multiple%20Doses%20Of%20GSI-953%20Within%20The%20Elderly%20Population